CLINICAL TRIAL: NCT06050915
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Single and Multiple Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity Characteristics of DISC-3405 in Adult Healthy Male and Female Volunteers
Brief Title: A Study of DISC-3405 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Disc Medicine, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DISC-3405-101
Record Dates: First submitted 2023-09-07; First posted 2023-09-22 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Single Ascending Dose of DISC-3405 (Experimental)
  Interventions: Drug: DISC-3405
- Single Ascending Dose of Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Multiple Ascending Dose of DISC-3405 (Experimental)
  Interventions: Drug: DISC-3405
- Multiple Ascending Dose of Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DISC-3405 — DISC-3405 is administered as a single dose IV infusion or subcutaneous injection
  Other Names: 9MW3011
  Arms: Single Ascending Dose of DISC-3405
Drug: DISC-3405 — DISC-3405 is administered in multiple ascending doses as an IV infusion or subcutaneous injection
  Other Names: 9MW3011
  Arms: Multiple Ascending Dose of DISC-3405
Drug: Placebo — Placebo is administered as a single dose IV infusion or subcutaneous injection
  Arms: Single Ascending Dose of Placebo
Drug: Placebo — Placebo is administered in multiple ascending doses as an IV infusion or subcutaneous injection
  Arms: Multiple Ascending Dose of Placebo

SUMMARY:
This phase 1 study will assess the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of DISC-3405 in adult male and female healthy volunteers.

DETAILED DESCRIPTION:
Each enrolled subject will receive one single or multiple doses of DISC-3405 or placebo. During the study, subjects will be evaluated for safety and tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of DISC-3405. In the single ascending dose (SAD) phase, a sentinel group of two subjects will be dosed first: one with DISC-3405, and the other with placebo; the randomization and blinding will be maintained. The remaining subjects for the cohort will be dosed at least 24 hours after the last sentinel dosing following approval from the principal investigator.

Subsequent multiple ascending dose (MAD) cohorts will only enroll after a sufficient safety observation period for the SAD cohort, accordingly there will be no sentinel participants for cohorts in MAD.

DISC-3405 or placebo will be administered as an IV infusion or subcutaneous injection. Subjects will have end-of-study (EOS) follow-up visits on Day 99 after the last administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, non-smokers, ages 18-65 (inclusive) at the time of signing the informed consent
* No clinically significant medical history and in good health as determined by detailed medical history
* Body mass index (BMI) 18.0 - 33.0 kg/m2 (inclusive) and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females

Exclusion Criteria:

* History of severe infection within 4 weeks prior to administration; signs and symptoms of any active infection regardless of severity within 2 weeks prior to administration.
* History of hypersensitivity to similar drugs to DISC-3405 or their excipients.
* Use of any prescription drugs, herbal supplements, or nonprescription drugs, including oral anti-histamines (for seasonal allergies), within 1 month or 5 half-lives (whichever is longer) prior to study drug administration, or dietary supplements within 1 week prior to study drug administration, unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study. Over-the-counter multivitamins will not be permitted. If needed, paracetamol/acetaminophen (up to 2 grams daily) may be used but must be documented in the Concomitant medications/Significant non-drug therapies page of the source data. Any questions of concomitant medications should be directed to the Sponsor.
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
* Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing
* Pregnant, or nursing females.
* A history of clinically significant psychiatric and psychological condition that, in the judgment of the investigator, may interfere with the planned treatment and follow-up, affect subject compliance, or place the subject at high risk from treatment-related complications
* Abnormal and clinically significant ECG (QT-interval corrected according to Fridericia's formula [QTcF] > 450 msec).
* Clinically significant abnormal vital signs at screening (systolic blood pressure [SBP] <90 mmHg or ≥140 mmHg; diastolic blood pressure [DBP] <50 mmHg or ≥90 mmHg; heart rate <50 beats per minute [bpm] or >100 bpm).
* Clinically significant abnormal laboratory test results or positive serology test results for hepatitis b surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody at screening.
* Immunization with a live or attenuated vaccine is prohibited within 4 weeks prior to study drug administration. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) or live attenuated vaccines and are not allowed.
* Receipt of an immunoglobulin or blood product 90 days prior to dosing
* History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit [more than 7 units for women or 14 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%)] or taking a product containing alcohol 2 days prior to dosing, or positive alcohol breath test at screening.
* History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs [such as cocaine, phencyclidine (PCP), crack, opioid derivatives including heroin, and amphetamine derivatives] within 1 year prior to screening.
* Positive urine drug screen, including a cotinine test at screening and on Day -1.
* Active infection with COVID-19. Subjects who have quarantined and are no longer deemed infectious may enroll. Subjects who received a COVID-19 vaccine within 4 weeks prior to dosing, or plan to receive COVID-19 vaccine during the time of their study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 99 days
Incidence of treatment-emergent clinically abnormal physical exam | up to 99 days
Incidence of treatment-emergent clinically significant laboratory test results | up to 99 days
Incidence of treatment-emergent clinically significant electrocardiograms (ECGs) | up to 99 days
Incidence of treatment-emergent clinically abnormal vital signs | up to 99 days

SECONDARY OUTCOMES:
Plasma maximum measured drug concentration (Cmax) | up to 99 days
Time of maximum concentration (Tmax) | up to 99 days
Area under the concentration-time curve from dosing to the last measurable time point (AUC0-t) | up to 99 days
Area under the concentration-time curve from dosing to infinity (AUC0-∞) | up to 99 days
Drug elimination half-life (T½ el) | up to 99 days
Volume of plasma cleared (CL) | up to 99 days
Trough Concentration (Ctrough) | up to 99 days
Volume of Distribution (Vd) | up to 99 days
Elimination rate constant (Kel) | up to 99 days
Change from baseline of hepcidin levels | up to 99 days
Change from baseline in transferrin saturation (TSAT) levels | up to 99 days
Change from baseline of serum iron levels | up to 99 days

CONTACTS AND LOCATIONS:
Overall Officials: Will Savage, MD PhD, Study Director — Disc Medicine
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No